CLINICAL TRIAL: NCT02575378
Title: Maintenance Treatment With Capecitabine Metronomic Chemotherapy and Chinese Traditional Medicine in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hao Li, associate chief physician, Department of Oncology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHYY-ZYYZX-rjzl
Record Dates: First submitted 2015-10-10; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Maintenance Treatment; Chinese Traditional Medicine; Clinical Trial; efficacy; safety
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronomic chemotherapy (Other): Metronomic Chemotherapy for maintenance treatment with Capecitabine 300mg/m2 twice a day, everyday.
  Interventions: Drug: Metronimic chemotherapy
- Metronimic chemotherapy plus Chinese Traditional Medicine (Experimental): Metronomic Chemotherapy for maintenance treatment with Capecitabine 300mg/m2 twice a day, everyday.
  Chinese Traditional Medicine
  Interventions: Drug: Metronimic chemotherapy plus Chinese Traditional Medicine

INTERVENTIONS:
Drug: Metronimic chemotherapy plus Chinese Traditional Medicine — Capecitabine 300mg/m2, twice a day, everyday plus Chinese Traditional Medicine
  Arms: Metronimic chemotherapy plus Chinese Traditional Medicine
Drug: Metronimic chemotherapy — Capecitabine 300mg/m2, twice a day, everyday
  Arms: Metronomic chemotherapy

SUMMARY:
The optimum regimen of maintenance treatment after first-line chemotherapy in patients with metastatic colorectal cancer （mCRC） is unknown. This study was designed to determine the efficacy and safety of maintenance treatment with capecitabine metronomic chemotherapy plus Chinese Traditional Medicine.

In this Prospective, open-label, randomised controlled trial, the investigators will recruit 159 mCRC patients who have finished 18 to 24 weeks first-line chemotherapy and disease evaluation is SD, PR or CR. The patients will then accept Chinese traditional diagnosis and be randomised into two group, capecitabine metronomic chemotherapy only as control group and the metronomic chemotherapy plus Chinese Traditional Medicine as experimental group. This treatment regimen will be continued until progression, death, or an unacceptable adverse event.

The primary endpoint is progression-free survival (PFS). Secondary endpoints are overall survival (OS), quality of life (QOL) and toxic effects.

ELIGIBILITY:
Inclusion Criteria:

1. unresectable metastatic colorectal cancer with pathological confirmation.
2. patients have accepted 18-24 weeks first-line chemotherapy and disease evaluation is SD, PR or CR.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | six months
  from randomising to progression, death, unacceptable AE